CLINICAL TRIAL: NCT03177980
Title: Fentanyl and Clonidine for Analgesia During Hypothermia in Term Asphyxiated Infants - a Prospective Pharmacokinetic/Pharmacodynamic/Pharmacogenetic Observational Study. Cohort 1 in The SANNI Project.
Brief Title: Fentanyl and Clonidine for Analgesia During Hypothermia in Term Asphyxiated Infants
Acronym: SANNI 1
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Karolinska Institutet (Other); Helsinki University Central Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Örebro University, Sweden (Other); The Swedish Research Council (Other Government); University of Colorado, Denver (Other); University of Tartu (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-002470-20
Record Dates: First submitted 2017-04-21; First posted 2017-06-06 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Asphyxia Neonatorum
Keywords: Term infants; Analgesia; fentanyl; clonidine; pharmacokinetics; sedation; pharmacodynamics; neurophysiology; pharmacogenetics; asphyxia; hypothermia
MeSH Terms: conditions — Asphyxia Neonatorum; Agnosia; Asphyxia; Hypothermia | interventions — Fentanyl; Clonidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fentanyl: All infants in need of analgesia according to an algorithm based on pain assessment results will receive fentanyl as the first analgesic drug.
  Interventions: Drug: Fentanyl
- Fentanyl and Clonidine: Infants in need of further analgesia according to an algorithm based on pain assessment results will receive fentanyl and clonidine as the analgesic drugs.
  Interventions: Drug: Fentanyl and clonidine

INTERVENTIONS:
Drug: Fentanyl — The dosing and administration of fentanyl will serve as the first drug intervention in infants in need of analgesia according to an algorithm based on pain scoring results.
  Groups: Fentanyl
Drug: Fentanyl and clonidine — In infants in need of further analgesia clonidine will be administered as an add on drug according to an algorithm based on pain scoring results.
  Groups: Fentanyl and Clonidine

SUMMARY:
A prospective pharmacokinetic (PK), pharmacodynamic (PD) and pharmacogenetic (PG) observation study, including the PK/PD/PG relationship, in fentanyl and clonidine administered for analgesia and sedation to term newborn asphyxiated infants receiving hypothermic treatment in the NICU.

DETAILED DESCRIPTION:
All patients that are admitted to the study neonatal intensive care units (NICUs) for hypothermic treatment due to perinatal asphyxia are potential study patients, and their parents will be asked for consent.

The patient will be treated according to clinical guidelines and will be included in the study if in need for fentanyl and clonidine according to clinical judgment (HIE and pain scores) and as decided by the responsible clinical doctor. The dosing and administration of the drugs will be implemented according to an algorithm based on pain scoring results.

Apart from extra blood sampling, the bedside monitoring, investigations (electroencephalography (EEG), echocardiography (ECG), ultrasound of the brain and magnetic resonance imaging, (MRI)) and follow-up (neurologic examination) are the same as for all infants receiving hypothermia according to national and international guidelines. A brief standardised pain stimulation will be performed as part of the pain and stress assessment.

In total 50 infants will be included.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (≥ gw 36+0) who, according to national guidelines (6), will receive hypothermic treatment following perinatal asphyxia, and are in need for analgesic or sedative medication according to clinical judgment based on Thomsons score and ALPS-Neo.
* Existing arterial or venous cannulas/catheters for repeated non-traumatic blood sampling
* Informed and written parental consent.

Exclusion Criteria:

* Atrioventricular (AV)- block I-III or heart rate < 70 .
* Serious coronary heart disease with need for postnatal surgery
* Mean arterial blood pressure <35 mmHg despite adequate treatment.

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Term asphyxiated infants admitted to the NICU for hypothermic treatment according to national and international guidelines and in need for analgesia according to pain assessment scales.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of fentanyl and clonidine | Repeated blood samples over a total of 4 - 7 days]
  Analysed with NONMEM (Non-linear Mixed Effect Modelling) populationbased PK statistics
Neurophysiologic response; by single cortical events and their dynamics in relation to PK | From admission to the department until 4- 72 h after reaching normothermia.]
  Analyse of single cortical events and their dynamics based on burst detection and measuring features of individual bursts as well as their mass statistical behaviour over time.
Neurophysiologic response; longer term brain function in relation to PK | From admission to the department until 4- 72 h after reaching normothermia
  Assessment of longer term brain function using measures of long range correlation and brain activity cycling.
Neurophysiologic response; global brain network function in relation to PK | From admission to the department until 4- 72 h after reaching normothermia
  Assessment of global brain network function will be based on Activation Synchrony Index.

SECONDARY OUTCOMES:
Change in/association between physiological parameters (heart rate, blood pressure, peripheral oxygen saturation and NIRS (near-infrared reflectance spectroscopy near-infrared spectroscopy) parameters) in relation to PK parameters | From admission to the department until 4- 72 h after reaching normothermia.
Change in pain responses as measured by pain assessment score for continuous pain/stress (ALPS-Neo and Comfort Neo) in relation to PK | From admission to the department until 4- 72 h after reaching normothermia.
Procedural pain response at a short standardized pain stimulation; as assessed with change in galvanic skin response, change in serum-cortisol and scored by a procedural pain assessment scale (PIPP-R) in relation to PK. | Once during stable treatment with hypothermia and 6 hours of unchanged medication
Pharmacogenetic profile in relation to PK and PD results; how PK/PD phenotypes depend on pharmacogenetic (PG) profiles. | One blood sample during study

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Norman, MD, Principal Investigator — Region Skane and Lunds University
Locations (2):
- Sweden (2):
  - Skåne Uniersity Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No